CLINICAL TRIAL: NCT06889688
Title: A Multicenter, Phase III, Randomized Controlled Trial Comparing Camrelizumab Plus Apatinib and Eribulin Versus Physician's Choice Chemotherapy in the Treatment of Advanced Triple-Negative Breast Cancer
Brief Title: Phase III Trial of Camrelizumab+Apatinib+Eribulin vs. Physician's Choice Chemotherapy in Advanced Triple-Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Jieqiong Liu, M.D., Ph.D., Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPER-III
Record Dates: First submitted 2025-03-11; First posted 2025-03-21 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Camrelizumab (200 mg, IV, Day 1) + Apatinib (250 mg, PO, QD) + Eribulin (1.4 mg/m², IV, Day 1 and Day 8) administered in 21-day cycles.
  Interventions: Drug: Camrelizumab+Apatinib+Eribulin
- Control Group (Active Comparator): Physician's Choice Chemotherapy
  Interventions: Drug: Physician's choice chemotherapy

INTERVENTIONS:
Drug: Camrelizumab+Apatinib+Eribulin — Camrelizumab (200 mg, IV, Day 1) + Apatinib (250 mg, PO, QD) + Eribulin (1.4 mg/m², IV, Day 1 and Day 8) administered in 21-day cycles.
  Arms: Experimental Group
Drug: Physician's choice chemotherapy — Physician's Choice Chemotherapy
  Arms: Control Group

SUMMARY:
This study evaluates the efficacy and safety of camrelizumab, apatinib, and eribulin versus physician's choice chemotherapy in advanced TNBC.Primary Objectives: Assess improvements in progression-free survival (PFS) and overall survival (OS).Secondary Objectives: Compare objective response rate (ORR), disease control rate (DCR), clinical benefit rate (CBR), duration of response (DoR), time to response (TTR), two-year OS rate, biomarker analysis, and quality of life (QoL).Safety: Assess and compare adverse event incidence and severity.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of the triplet regimen compared to physician's choice chemotherapy as a later-line treatment for advanced triple-negative breast cancer (TNBC). 1. Primary Objectives and Endpoints: To determine whether the combination of camrelizumab, apatinib, and eribulin improves progression-free survival (PFS) and overall survival (OS) compared to investigator's choice chemotherapy in advanced TNBC. 2. Secondary Objectives and Endpoints: To compare the following clinical parameters between the camrelizumab, apatinib, and eribulin combination and investigator's choice chemotherapy for advanced TNBC: -Objective response rate (ORR) Disease control rate (DCR) Clinical benefit rate (CBR) Duration of response (DoR) Time to response (TTR) Two-year overall survival rate (2-year OS rate) Biomarker analysis Quality of life (QoL) analysis 3.Safety Evaluation: Comparison of the incidence and severity of adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily agrees to participate in this study and signs an informed consent form (ICF).
2. Female subjects aged ≥18 and ≤70 years on the date of signing the ICF.
3. Pathologically confirmed advanced triple-negative breast cancer (TNBC), defined as ER-negative (IHC ER-positive percentage <1%), PR-negative (IHC PR-positive percentage <1%), and HER2-negative (IHC-/+, or IHC++ but FISH/CISH-), with at least one measurable lesion per RECIST v1.1 criteria.
4. Previously received ≥1 line of systemic therapy for metastatic or locally advanced unresectable TNBC with disease progression. Prior systemic therapy (including ≥1 line of chemotherapy and neoadjuvant/adjuvant chemotherapy) must have included a taxane or anthracycline. Recurrence within 6 months after completing neoadjuvant/adjuvant chemotherapy is considered as failure of first-line therapy.
5. Capable of swallowing tablets.
6. ECOG performance status of 0-1.
7. Expected survival ≥12 weeks.
8. Adequate function of vital organs, meeting the following criteria (without the use of blood products or growth factors during the screening period): Absolute neutrophil count (ANC) ≥1.5×10⁹/L. Platelet count ≥100×10⁹/L. Hemoglobin ≥9 g/dL. Serum albumin ≥3 g/dL. Thyroid-stimulating hormone (TSH) ≤ULN (if abnormal, T3 and T4 levels should be assessed; subjects with normal T3 and T4 levels are eligible). Total bilirubin ≤1.0×ULN (for subjects with Gilbert's syndrome or liver metastases, total bilirubin ≤1.5×ULN). ALT and AST ≤1.5×ULN (for subjects with liver metastases, ≤3×ULN). Alkaline phosphatase (ALP) ≤2.5×ULN. Renal function within 7 days prior to the first dose: serum creatinine ≤1.5×ULN or creatinine clearance ≥60 mL/min.
9. Women of childbearing potential agree to use highly effective contraception starting at least 7 days prior to the first dose and continuing for 24 weeks after the last dose. A negative serum pregnancy test is required within 7 days prior to the first dose.

Exclusion Criteria:

1. Subjects with untreated active brain metastases or leptomeningeal metastases.
2. Participation in any other interventional clinical trial within 28 days prior to the first dose.
3. History of severe allergic reactions to other monoclonal antibodies.
4. Receipt of other antitumor therapies within 28 days prior to the first dose.
5. Uncontrolled hypertension despite antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg).
6. Prior treatment with CTLA-4, Tim-3, or LAG-3 antibodies, or T-cell co-stimulatory therapies (previous use of PD-1 or PD-L1 antibodies is allowed).
7. Prior treatment with anti-angiogenic agents or eribulin chemotherapy.
8. Presence of any active autoimmune disease or a history of autoimmune disease (including but not limited to autoimmune hepatitis, interstitial pneumonitis, uveitis, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, or hypothyroidism). Subjects with vitiligo, or childhood asthma that has fully resolved without intervention in adulthood, may be included. Subjects with asthma requiring medical intervention with bronchodilators are excluded.
9. Uncontrolled cardiac clinical symptoms or diseases, including: Heart failure classified as NYHA Class II or higher. Unstable angina. Myocardial infarction within the past year. Clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention.
10. Urinalysis indicating proteinuria ≥++ or confirmed 24-hour urinary protein ≥1.0 g.
11. Known hereditary or acquired bleeding or thrombotic disorders (e.g., hemophilia, coagulopathy, thrombocytopenia, hypersplenism).
12. Congenital or acquired immunodeficiency (e.g., HIV infection).
13. Receipt of a live vaccine within 4 weeks prior to or during the study period.
14. Allergy or contraindication to the investigational drugs.
15. Underwent surgery within 3 months prior to enrollment or anticipated need for major surgical procedures during the study period.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2030-09-20 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Time from enrollment to the occurrence of predefined events, including disease progression or death, whichever came first, assessed up to 60 months.
  Disease evaluation will be performed according to RECIST v1.1 criteria.
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 120 months.
  Death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented CR or PR, whichever came first, assessed up to 12 months.
  The percentage of patients in different groups whose tumor size reduction, meets the criteria for complete response (CR) or partial response (PR).
Disease control rate | From date of randomization until the date of first documented CR, PR or SD, assessed up to 12 months.
  Proportion of patients achieving CR, PR, or stable disease (SD).
Clinical Benefit Rate | From date of randomization until the date of first documented CR, PR or SD for more than 6month, assessed up to 18 months.
  Proportion of patients achieving CR, PR, or SD.
Duration of Response | Time from the first assessment showing CR or PR to the first occurrence of PD or death from any cause, whichever came first, assessed up to 120 months.
  Time from the first assessment showing CR or PR to the first occurrence of progressive disease (PD) or death from any cause.
Time to Response | Time from randomization to the first occurrence of CR or PR, whichever came first, assessed up to 6 months
  Time from randomization to the first occurrence of CR or PR.
Two-Year Overall Survival Rate | Two years after randomization.
  Proportion of patients alive two years after randomization.
Safety Evaluation | From randomization to 30 days after the last dose of study treatment.
  Comparison of the incidence and severity of adverse events between the two groups.

OTHER OUTCOMES:
Tumor and Peripheral Blood Biomarker Analysis | Before treatment and after 2 cycles (each cycle is 21 days) of treatment, or disease progression.
  This analysis aims to identify biomarkers that predict treatment response, resistance, and prognosis in advanced triple-negative breast cancer (TNBC).
  Tumor Biomarker Analysis:
  Genetic and Molecular Profiling: Whole-exome sequencing (WES), RNA sequencing, and proteomics to identify mutations, gene expression patterns, and protein markers related to treatment response.
  Immune Microenvironment Assessment: Immunohistochemistry (IHC) and multiplex immunofluorescence to evaluate tumor-infiltrating lymphocytes (TILs), PD-L1 expression, and other immune-related markers.
  Peripheral Blood Biomarker Analysis: Measurement of inflammatory and immunomodulatory cytokines to assess systemic immune response.
QoL | At baseline upon enrollment and every 2cycles (each cycle is 21 days) of treatment, from date of randomization until the patient exits the study due to disease progression, adverse events, whichever came first, assessed up to 60 months.
  Quality of life assessment will be conducted using the EORTC QLQ-BR23 questionnaire. Raw scores will be linearly transformed to a standardized scale ranging from 0 to 100 points.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Wuhan Union Hospital of China, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - The Central Hospital Of Yong Zhou, Yongzhou, Hunan

IPD SHARING:
Plan to Share IPD: No